CLINICAL TRIAL: NCT03876223
Title: Women's Ischemia Syndrome Evaluation (WISE) Mechanisms of Coronary Microvascular Dysfunction Leading to Pre-Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Women's Ischemia Syndrome Evaluation (WISE) Pre-HFpEF
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Other Study IDs: 54999
Record Dates: First submitted 2019-02-22; First posted 2019-03-15 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Coronary Microvascular Dysfunction; Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: Coronary Microvascular Dysfunction (CMD); Coronary Vascular Dysfunction (CVD); Coronary angiography; Magnetic resonance imaging (MRI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A maximum of 45 mL of whole blood will be collected, which will be processed and stored as serum, plasma, and DNA for biomarkers and for genetic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to examine small vessel disease (a condition in which the small arteries in the heart become narrowed). The investigators want to know how the small vessel disease contributes to pre-HFpEF (a condition with inadequate heart muscle function in the setting of preserved muscle pumping) and to better identify potential treatment for prevention of HFpEF. The main procedures of this study include up to 2 clinic visits (initial visit and a second clinical visit only if participants are unable to complete all research procedures at the initial visit); a 6-week phone interview visit, 4 quarterly follow-up phone interview visits in year 1; year 1 follow up cardiac MRI based on availability and ongoing annual follow-up phone interview visits to track progress. If participants choose to take part in this study, participants direct participation will end after 1 year, participants will then have the option of participating in ongoing annual check-in calls. Participants will be asked to undergo a physical exam and provide a completed medical history; complete a Cardiovascular (or Cardiac) Magnetic Resonance Imaging (CMRI) with contrast agent; complete questionnaires to describe heart symptoms and overall quality of life status; undergo blood draws to provide blood samples for research testing, and allow the study team to have access to medical records.

DETAILED DESCRIPTION:
Coronary microvascular dysfunction (CMD) due to changes in the function and structure of coronary microcirculation in the absence of obstructive coronary artery disease (CAD) is poorly understood. Ischemia with no obstructive CAD (INOCA) and myocardial infarction with no obstructive CAD (MINOCA) are increasingly observed in women and men.

Once established, the investigators will be well positioned to aggressively target identified mechanistic targets in a specific well-characterized at-risk population, with the primary goal of preventing progression to HFpEF.

To address this novel hypothesis, the investigators propose the following Specific Aims:

Aim 1: Test the hypothesis that CMD-related ischemia contributes to myocellular damage and impaired ventricular relaxation. CMD will be measured directly, using our established intracoronary pharmacological vasoactive protocol, in subjects with signs/symptoms of ischemia but no obstructive CAD. In our labs (>420 patients), ~60% of those tested have evidence for CMD. All subjects will perform provocative stress testing with isometric handgrip - chosen for its unique ability to increase myocardial afterload and myocardial oxygen demand - while myocardial ischemia will be assessed directly through invasive simultaneous arterial and coronary sinus/great cardiac vein oxygen tension and lactate measurements, and continuous ECG's recordings. Left ventricular function will be directly assessed using Millar-catheter LV pressure-volume loops (perfected in our lab over the past 24 months). Stress-induced myocellular damage will be directly measured by coronary sinus/great cardiac vein hs-cTnI.

Aim 2: Test the hypothesis that CMD-related ischemic myocellular damage contributes to LV diastolic dysfunction progression. Subjects from Aim 1 will also undergo comprehensive cardiac magnetic resonance imaging (CMRI) at enrollment and 1-2 years later. The investigators will evaluate CMRI LV perfusion, myocardial scar, diffuse fibrosis, LV remodeling, and diastolic function. The investigatorswill leverage the strengths and resources of our world-renowned proteomics core to establish evidence of chronic myocellular damage using prospectively repeated ambulatory hs-cTnI determinations.

ELIGIBILITY:
Inclusion:

1. 180 symptomatic men and women undergoing invasive coronary angiography for suspected ischemia with no obstructive CAD, defined as ≥50% luminal diameter stenosis in ≥1 epicardial coronary artery.
2. Preserved left ventricular ejection fraction (EF) ≥45%
3. Be > 18 years old
4. Be able to meet the requirement for a cardiac MRI, which means no metal devices in your chest, no claustrophobia and no angioedema
5. Be competent to give informed consent

Exclusion:

1. Subjects with severe or chronic kidney disease (CKD) with GFR<405 or acute kidney injury
2. Subjects with allergy to animal dander will be excluded since imaging will be done in BIRI (BIRI scanners are also used to image animals).
3. Subjects who have had four or more prior previous gadolinium contrast scans
4. Allergy/ hypersensitivity to adenosine, gadolinium, aminophylline or regadenoson
5. Second- or third-degree A-V block
6. Sinus node disease, such as sick sinus syndrome or symptomatic bradycardia (except in patients with a functioning artificial pacemaker)
7. Subjects with mild to severe asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women undergoing invasive coronary angiography for suspected ischemia with no obstructive CAD, defined as ≥ 50% luminal diameter stenosis in ≥ 1 epicardial coronary artery.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
CMR imaging | Baseline, Annual follow up
  Change from Baseline at 1 year follow up will be assessed.
Rest-stress Millar pressure-volume measurement | Baseline
  LV diastolic function will be measured using LV end-diastolic pressure, minimal rate of LV pressure change (dP/dtmin).

SECONDARY OUTCOMES:
Questionnaire | Baseline, 6 week, quarterly(year 1) and annual follow up
  Symptom History Questionnaire. Change from Baseline at each visit will be measure. There is no scale ranges for this questionnaire. This questionnaire results in raw data that is not calculated into a score or scale.
Questionnaire WISE Symptoms History | Baseline, quarterly(year 1) and annual follow up
  Detailed information on chest pain symptoms will include the WISE female angina questionnaire.
  Change from Baseline at each visit will be measure. There is no scale ranges for this questionnaire. This questionnaire results in raw data that is not calculated into a score or scale.
SEATTLE ANGINA QUESTIONNAIRE | Baseline, 6 week and annual follow up
  The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life.
  Each scale is transformed to a score of 0 to 100. A higher score means better control of chest pain, chest tightness, angina, or shortness of breath.
  Change from Baseline at each visits will be measure.
Duke Activity Status Inventory (DASI) | Baseline, 6 week and annual follow up
  It is a self-administered questionnaire that measures a patient's functional capacity.
  Change from Baseline at each visit will be measure. Maximum response is a total of 16.7 while minimum is 0.

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, FACC, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Takahashi T, Wei J, Iribarren AC, Gulati M, Cook-Wiens G, Nelson MD, Sharif B, Handberg EM, Anderson RD, Petersen J, Berman DS, Pepine CJ, Merz CNB. Rationale and design of the women's ischemia syndrome evaluation mechanisms of coronary microvascular dysfunction leading to preheart failure with preserved ejection fraction (WISE Pre-HFPEF). Am Heart J. 2025 Jun;284:47-56. doi: 10.1016/j.ahj.2025.02.017. Epub 2025 Feb 24. PMID 40010584